CLINICAL TRIAL: NCT03861858
Title: Dialectical Behavior Therapy for Adolescents at Rutgers University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shireen L. Rizvi, PhD, ABPP, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018001563
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Borderline Personality Disorder in Adolescence
Keywords: borderline personality disorder; adolescence; suicide; substance use
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBT-A (Experimental): The standard treatment to be delivered to all participants is DBT-A, which is a treatment model adapted from DBT. DBT-A is an adaptation for adolescents with emotion dysregulation and BPD features (Miller, Rathus, & Linehan, 2007; Rathus & Miller, 2015). DBT-A involves weekly individual therapy with the adolescent, weekly multifamily skills group in which adolescents and family members participate, as needed phone coaching, and weekly consultation team for the therapists.
  Interventions: Behavioral: DBT-A

INTERVENTIONS:
Behavioral: DBT-A — DBT-A is a multimodal therapy which consists of weekly individual therapy, weekly multifamily skills groups, as needed phone coaching, and weekly consultation team for the therapists.

SUMMARY:
This project expands our existing psychological services clinic (the Dialectical Behavior Therapy Clinic at Rutgers University; DBT-RU) to include an adolescent treatment arm. Adolescents aged 13-20 and at least one caregiver will be recruited to participate in a six-month treatment study. Adolescents will be eligible to participate if they meet at least 3 criteria for borderline personality disorder, with one of those criteria being either impulsive behavior or recurrent self-harm behavior. Participants will be assessed at baseline, three-months (mid-treatment), six-months (post-treatment, and three-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 years or 18-20 if still living at home with parent.
* Agreement of at least one responsible adult parent/caregiver to participate in treatment.
* Agreement to take part in assessments, videotaping/audiotaping and coding of their sessions by research personnel.
* Agreement to pay for mental health services at the DBT- RU on a sliding scale, and to participate in research assessments as volunteers.
* Residence within commuting distance of clinic (< 45 minutes).
* Agreement to discontinue other forms of talk therapy for duration of DBT program (does not refer to AA/NA programs or psychotropic medication management).
* Exhibits dysregulation within the past six months as evidenced by 1) intentional self-injury and/or suicide attempt and/or 2) substance use disorder.
* Meets two additional criteria for borderline personality disorder (BPD).

Exclusion Criteria:

* Clients who need mental health services not available at the DBT- RU, such as treatment for schizophrenia or life-threatening anorexia, or who are currently obtaining optimum professional treatment that should not be ended.
* Non-English speaking.
* IQ < 70.
* Unable to understand research consent forms.
* Court-ordered to participate in treatment.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Self-Injurious Thoughts and Behaviors Inventory (SITBI) | six months
  semi-structured interview designed to assess presence of suicide ideation, suicide attempts, self-injurious behaviors
Work and Social Adjustment Scale | six months
  WSAS items are rated on a scale of 0 (No Impairment) to 8 (Severe Impairment). Total scores are calculated by adding the scores of all 5 items. The minimum score of the WSAS is 0 and the maximum score of the WSAS is 40. Scores below 10 are associated with subclinical populations. Scores between 10 and 20 are associated with significant impairment, but less severe clinical symptomology. Scores above 20 are associated with moderately severe or worse psychopathology.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | six months
  The DERS is a 36-item measure of the six facets of emotion regulation.
  DERS items are rated on a scale of 1 (Almost Never 0-10%) to 5 (Almost Always 91-100%). The DERS total score ranges from 36-180. The total score is the sum of all subscales. Higher scores suggest greater problems with emotion regulation.
Borderline Symptom List (BSL-23) | six months
  The BSL is a 23-item measure that assesses specific symptoms of borderline personality disorder.
  BSL items are measured on a scale of 0 (Not at all) to 4 (Very strong). The sum of all 23 items serves as the global scale factor. The global factor minimum score of the BSL is 0 and the maximum score is 92. To generate scores that are comparable to the original BSL-95, the mean score must be calculated. Higher total scores are associated with more symptoms of borderline personality disorder.
Brief Symptom Inventory (BSI) | six months
  The BSI is a 53-item measure of psychological distress and psychological symptoms.
  BSI items are rated on a scale from 0 (Not at all) to 5 (Extremely). The BSI consists of 9 symptom dimensions and 3 global indices of stress. All 9 dimensions (Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism) have a score range from 0-5. Dimension scores are calculated by summing the values for the items included in that dimension and dividing by the number of items endorsed in that dimension.
  The 3 global indices of stress are Global Severity Index, Positive Symptom Total, and Positive Symptom Distress Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No